CLINICAL TRIAL: NCT06538233
Title: A Comparison of Pain Response During Administration of Buffered Articaine Versus Non-buffered Articaine Local Anesthetics for Dental Treatment in Adult
Brief Title: Pain After Buffered Vs Non Buffered Articaine
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cleveland Dental Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDIOS00010
Record Dates: First submitted 2024-07-17; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buffered articaine (Experimental)
  Interventions: Drug: Buffered articaine
- non buffered articaine (Active Comparator)
  Interventions: Drug: Non buffered articaine

INTERVENTIONS:
Drug: Buffered articaine — Injecting buffered articaine in maxillary anterior region and evaluate pain response.
  Arms: Buffered articaine
Drug: Non buffered articaine — Injecting non buffered articaine in maxillary anterior region and evaluate pain response.
  Arms: non buffered articaine

SUMMARY:
Pain after buffered versus non buffered articaine.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age- 18 to 60 yrs.
* Medically free.
* Need a dental treatment in the upper anterior region.

Exclusion Criteria:

* Periodontally affected teeth.
* Radiographic bone loss.
* Upnormal length of the teeth.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Numerical Rate Scale (NRS) | Immediate
  Pain during injection of buffered versus non-buffered articaine local anesthetic will be measured using NRS from 0 to 10, where 0 is no pain and 10 is the most unbearable pain .

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed H Khalifa, PhD, Study Chair — Cleveland Dental Institute; Waleed Elmallah, PhD, Principal Investigator — Cleveland Dental Institute
Locations (1):
- Clevland Dental Institute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No